CLINICAL TRIAL: NCT07288034
Title: Immunotherapy Biomarker Collection for Metastatic NSCLC to Inform Adaptive Personalized Models Targeting Resistance (IMMUNO-BIOMAP)
Brief Title: Immunotherapy Biomarkers to Predict First-line PD(L)1-based Immunotherapy Response and Selection of Second-line Treatment in Stage IIIB-IV Non-small Cell Lung Cancer, IMMUNO-BIOMAP Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24507; NCI-2025-09032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24507 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — adagrasib; spartalizumab; Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; Drug Therapy; durvalumab; Magnetic Resonance Spectroscopy; tremelimumab

STUDY DESIGN:
Intervention Model Description: Randomized Part IA, Future Part IB to replace Part IA, and a non-randomized Part II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1 (stop treatment, monitoring) (Experimental): Patients receive physician's choice of PD(L)1-based therapy Q3W with or without chemotherapy for up to 12-24 months per standard of care. After at least 12 months of treatment, patients discontinue PD(L)1 therapy and undergo monitoring. Patients who develop positive ctDNA without PD resume PD(L)1 on study. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care and tumor biopsy throughout the study.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody; Biological: Anti-PD1 Monoclonal Antibody; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Monitoring; Procedure: Positron Emission Tomography
- Arm 2 (continue PD[L]1) (Experimental): Patients receive physician's choice of PD(L)1-based therapy Q3W with or without chemotherapy for up to 12-24 months per standard of care. After at least 12 months of treatment, patients continue PD(L)1 therapy for up to a total of 24 months from starting immunotherapy in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care and tumor biopsy throughout the study.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody; Biological: Anti-PD1 Monoclonal Antibody; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm 3 (close surveillance) (Experimental): Patients receive physician's choice of PD(L)1-based therapy Q3W with or without chemotherapy for up to 12-24 months per standard of care. After at least 24 months of treatment, patients discontinue PD(L)1 therapy and undergo close surveillance on study. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care and tumor biopsy throughout the study.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody; Biological: Anti-PD1 Monoclonal Antibody; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Behavioral: Surveillance
- Arm 4 (PD[L]1) (Experimental): Patients receive physician's choice of PD(L)1-based therapy Q3W with or without chemotherapy for up to 12-24 months per standard of care. After at least 24 months of treatment, patients continue to receive PD(L)1 therapy until radiographic progression or unacceptable toxicity. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care and tumor biopsy throughout the study.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody; Biological: Anti-PD1 Monoclonal Antibody; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm A (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV over 1 hour on day 1 of cycles 1-4 and on day 1 of cycle 6 as well as durvalumab IV over 1 hour of each cycle. Cycles repeat every 21 days for cycles 1-5 and then starting with cycle 6, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tremelimumab
- Arm B (adagrasib, bevacizumab) (Experimental): Patients receive adagrasib PO BID on days 1-21 and bevacizumab IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may undergo CSF, ascites and pleural fluid sample collection during routine care throughout the study.
  Interventions: Drug: Adagrasib; Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Adagrasib — Given PO
  Other Names: KRAS G12C Inhibitor MRTX849; Krazati; MRTX 849; MRTX-849; MRTX849
  Arms: Arm B (adagrasib, bevacizumab)
Biological: Anti-PD-L1 Monoclonal Antibody — Given PD-L1-based immunotherapy
  Arms: Arm 1 (stop treatment, monitoring); Arm 2 (continue PD[L]1); Arm 3 (close surveillance); Arm 4 (PD[L]1)
Biological: Anti-PD1 Monoclonal Antibody — Given PD1-based immunotherapy
  Other Names: Anti-PD-1 Monoclonal Antibody
  Arms: Arm 1 (stop treatment, monitoring); Arm 2 (continue PD[L]1); Arm 3 (close surveillance); Arm 4 (PD[L]1)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm B (adagrasib, bevacizumab)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm 1 (stop treatment, monitoring); Arm 2 (continue PD[L]1); Arm 3 (close surveillance); Arm 4 (PD[L]1)
Procedure: Biospecimen Collection — Undergo blood, CSF, ascites and pleural fluid sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Chemotherapy — Given chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Arm 1 (stop treatment, monitoring); Arm 2 (continue PD[L]1); Arm 3 (close surveillance); Arm 4 (PD[L]1)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm A (tremelimumab, durvalumab)
Procedure: Magnetic Resonance Imaging — Undergo PET
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Monitoring — Undergo monitoring
  Other Names: monitor
  Arms: Arm 1 (stop treatment, monitoring)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Behavioral: Surveillance — Undergo close surveillance
  Other Names: Epidemiology / Surveillance
  Arms: Arm 3 (close surveillance)
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP 675; CP 675206; CP-675; CP-675,206; CP-675206; CP675; CP675206; Imjudo; Ticilimumab; Tremelimumab-actl
  Arms: Arm A (tremelimumab, durvalumab)

SUMMARY:
This phase II trial tests the impact of biomarkers in predicting initial treatment (first-line) PD1 or PD-L1 (PD[L]-1)-based immunotherapy response and in selecting second-line treatment in patients with stage IIIB-IV non-small cell lung cancer (NSCLC). Response and survival rates in advanced stage NSCLC, unlike other cancers, rely on response to first-line therapy. Immunotherapy with PD(L)1-based therapy, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. While immunotherapy has improved survival rate, the prognosis remains poor with most patients receiving chemotherapy after immunotherapy. Many types of tumors tend to lose cells or release different types of cellular products including their deoxyribonucleic acid (DNA) which is referred to as circulating tumor DNA (ctDNA) into the bloodstream before changes can be seen on scans. Health care providers can measure the level of ctDNA in blood or other bodily fluids to determine which patients are at higher risk for disease progression or relapse. The first part of this trial, studying samples of blood and tissue in the laboratory from patients receiving immunotherapy may help doctors learn more about the effects PD(L)1-based therapy on cells. It may also help doctors understand how well patients respond to treatment and may help develop new individualized treatment strategies. The second part of this trial also tests the effect of second-line immunotherapy, such as tremelimumab and durvalumab or adagrasib and bevacizumab, in treating patients with NSCLC with specific genetic mutations that is growing, spreading or getting worse (progressive). Tremelimumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Adagrasib, a type of targeted therapy, may stop the growth of tumor cells by blocking a protein needed for tumor cell growth and may kill them. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Giving second-line immunotherapy, tremelimumab and durvalumab or adagrasib with bevacizumab, may be safe, tolerable, and/or effective in treating patients with stage IIIB/IV NSCLC with specific genetic mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop biomarker(s) that predicts for first-line treatment failure of immunotherapy (Part I).

II. Evaluate different strategies for treatment duration for patients without early treatment failure based on ctDNA (Part I).

III. Evaluate second-line progression-free survival (PFS) for biomarker-specific treatment decisions compared to historical controls (Part II).

SECONDARY OBJECTIVES:

I. Evaluate different ctDNA-guided treatment decisions on overall survival based on arm.

II. Summarize the relationship between ctDNA changes and Response Evaluation Criteria in Solid Tumors (RECIST) response throughout the trial.

III. To describe the incidence and severity of adverse events by treatment arm. IV. Demonstrate the feasibility of an adaptive design employing both dynamic treatment regimen and biomarker-specific directed therapy.

EXPLORATORY OBJECTIVE:

I. Use data from ctDNA and tissue multi-omics analysis for reverse translational modeling for mechanisms of resistance to immunotherapy using ARTEMIS.

OUTLINE:

PART IA (INITIAL DISCOVERY COHORT): Patients receive physician's choice of PD(L)1-based therapy every 3 weeks (Q3W) with or without chemotherapy for up to 12-24 months per standard of care.

Patients who complete at least 12 months of PD(L)1 (but do not exceed 24 months) and achieve complete response (CR), stable disease (SD), or partial response (PR) on imaging, as well as ctDNA complete response (CCR) for at least 6 months are randomized to Arms 1 or 2.

ARM 1: After at least 12 months of treatment, patients discontinue PD(L)1 therapy and undergo monitoring. Patients who develop positive ctDNA without PD resume PD(L)1 on study.

ARM 2: After at least 12 months of treatment, patients continue PD(L)1 therapy for up to a total of 24 months from starting immunotherapy the absence of disease progression or unacceptable toxicity.

Patients who complete 24 months of immunotherapy and achieve CR, SD, or PR on imaging, but not CCR and who were not candidates for Arms 1 and 2 are randomized to Arms 3 or 4.

ARM 3: After at least 24 months of treatment, patients discontinue PD(L)1 therapy and undergo close surveillance on study.

ARM 4: After at least 24 months of treatment, patients continue to receive PD(L)1 therapy until radiographic progression or unacceptable toxicity.

PART IB (IMPLEMENTATION COHORT): Patients participate in a future implementation cohort utilizing the findings from Part 1A.

PART II (POST-PROGRESSION COHORT): Patients who experience radiographic progression on Part I are assigned to 1 of 3 arms. Patients with STK11 or KEAP1 mutations are assigned to Arm A and patients with KRAS G12C mutations are assigned to Arm B. Patients assigned to Arm X will be added based on the funding grant technical area 1 (TA1-Therapy Recommendation Techniques).

ARM A: Patients receive tremelimumab intravenously (IV) over 1 hour on day 1 of cycles 1-4 and on day 1 of cycle 6, as well as durvalumab IV over 1 hour of each cycle. Cycles repeat every 21 days for cycles 1-5 and then starting with cycle 6, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive adagrasib orally (PO) twice daily (BID) on days 1-21 and bevacizumab IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM X: Patients participate in future interventions to be added based on the funding grant TA1-Therapy Recommendation Techniques.

Patients in both Parts also undergo blood sample collection, and computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET) throughout the study. Additionally, patients may undergo cerebrospinal fluid (CSF), ascites and pleural fluid sample collection during routine care throughout the study. Patients in Part 1 only undergo a tumor biopsy throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3 months within 1 year of starting treatment, then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative. (Adult patients lacking capacity to consent may participate if they have a caretaker that could ensure compliance.)
* Participants must have either A) HopeSeq or Tempus molecular testing results reported within 3 months prior to enrollment or currently in process OR B) archival or new biopsy tissue available (to be sent to Tempus). Acceptable sample types include: two formalin-fixed paraffin-embedded (FFPE) tissue core biopsies, or two 25um sections of 5-10mm^2 tissue, or 15-20 unstained slides at 10um thickness (a minimum of 10 unstained slides must be provided)
* Agreement to blood collection for ctDNA research
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed stage IIIB or IV NSCLC
* Absence of sensitizing EGFR mutation or ALK/ROS1 alteration
* Scheduled to begin treatment with a Food and Drug Administration (FDA) approved PD1/PDL1 antibody with or without chemotherapy. Participants who have already started treatment with anti-PD1/PDL1 in this setting may enroll if they have only received up to 4 cycles of treatment so far. Patients who have received PD1/PDL1 antibody for early-stage NSCLC are allowed to enroll if they completed the therapy at least 6 months before starting trial therapy
* Measurable disease by RECIST version (v) 1.1
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment
* Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment
* Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN (5 x ULN allowed if liver metastases)
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN (5 x ULN allowed if liver metastases)
* Creatinine clearance of ≥ 50 mL/min per the Cockcroft-Gault formula
* If seropositive for HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV), nucleic acid quantitation must be performed. Viral load must be undetectable

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* PART II: Documented informed consent (for Part II) of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* PART II: ECOG ≤ 2
* PART II: Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* PART II: ANC ≥ 1,500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment
* PART II: Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment
* PART II: Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment
* PART II: Total bilirubin ≤ 1.5 x ULN
* PART II: AST ≤ 3.0 x ULN (5 x ULN allowed if liver metastases)
* PART II: ALT ≤ 3.0 x ULN (5 x ULN allowed if liver metastases)
* PART II: Creatinine clearance of ≥ 50 mL/min per the Cockcroft-Gault formula

Exclusion Criteria:

* Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement
* Patients with a condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) within 7 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Radiation therapy within 7 days prior to day 1 of protocol therapy
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association [NYHA class] ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs
* Symptomatic central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have 1) previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug OR 2) untreated brain metastases that are asymptomatic and stable
* Prior history of interstitial lung disease (ILD) or non-infectious pneumonitis requiring high-dose glucocorticoids
* Active infection requiring antibiotics
* Other active malignancy. Patients with concurrent malignancy other than non-melanoma skin cancer are not eligible for this trial due to potential confounding of the ctDNA results
* Females only: Pregnant or breastfeeding
* PART II: Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement
* PART II: Radiation therapy within 7 days prior to day 1 of protocol therapy
* PART II ARM A ONLY: Patients with a condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) within 7 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* PART II ARM A ONLY: Patients with prior history of cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) treatment
* PART II ARM B ONLY: Patients with prior history of KRAS G12C inhibitors
* PART II: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication
* PART II ARM A ONLY: Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs
* PART II ARM B ONLY: Grade ≥ 2 proteinuria as demonstrated by ≥ 2+ protein and ≥ 1.0 g of protein with 24-hour urine collection (patients found to have ≥ 2+ protein on dipstick urinalysis must have 24-hour urine collection and demonstrate < 1g of protein in 24 hours in order to be eligible for treatment)
* PART II: Clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have 1) previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug OR 2) untreated brain metastases that are asymptomatic and stable
* PART II: Clinically significant uncontrolled illness
* PART II: Active infection requiring antibiotics
* PART II: Other active malignancy
* PART II FEMALES ONLY: Pregnant or breastfeeding
* PART II: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2026-09-21 (Estimated); Primary Completion 2028-09-22 (Estimated); Study Completion 2028-09-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) during first-line treatment (Part I) | From the start of randomization to disease progression or death from any cause, whichever occurs first, assessed up to 3 years
  Will be estimated using the Kaplan-Meier (KM) method. Comparisons across treatment arms will be performed using stratified log-rank tests and Cox proportional hazards models, with assessment of the proportional-hazards assumption and exploration of time-dependent hazard ratios. Dynamic treatment regimen (DTR)-specific PFS will also be estimated using inverse probability weighting (IPW) to account for multiple randomizations and treatment adaptations.
PFS by arm for second-line treatment (Part II) | From the start of treatment to disease progression or death from any cause, whichever occurs first, assessed up to 3 years
  Will be estimated using the KM method. Comparisons across treatment arms will be performed using stratified log-rank tests and Cox proportional hazards models, with assessment of the proportional-hazards assumption and exploration of time-dependent hazard ratios. DTR-specific PFS will also be estimated using IPW to account for multiple randomizations and treatment adaptations.

SECONDARY OUTCOMES:
Development and testing of biomarkers predictive of early response to immunotherapy | At pre-treatment and Cycle 2 Day 1 (blood only) (Cycle length = 21 days)
  Will include, but not limited to, blood based, tissue-based and imaging-based biomarkers.
Overall survival (OS) | From randomization (by arm and from start of first-line treatment) to death due to any cause, assessed up to 3 years
  Will be evaluated by arm. Will be estimated using the KM method. Comparisons across treatment arms will be performed using stratified log-rank tests and Cox proportional hazards models, with assessment of the proportional-hazards assumption and exploration of time-dependent hazard ratios. DTR-specific OS will also be estimated using IPW to account for multiple randomizations and treatment adaptations.
Circulating tumor deoxyribonucleic acid (ctDNA) level | Up to 3 years
  Joint modeling approaches will be applied, combining mixed-effects models for ctDNA trajectories with survival models for PFS or OS. All stratified efficacy analyses will incorporate randomization stratification factors.
ctDNA complete response (CCR) rate | Up to 3 years
  Will be summarized by treatment sequence. Logistic regression models will evaluate associations between CCR and baseline covariates.
Objective response rate (ORR) | From start of the study treatment to disease progression or death due to any cause prior to receiving another therapy, whichever occurs first, assessed up to 3 years
  Will be defined as rate of participants achieving confirmed complete response or partial response, as assessed by the investigator using Response Evaluation Criteria in Solid Tumors version (v) 1.1. ORR point estimates and 95% confidence intervals will be calculated using Clopper-Pearson methods, and logistic regression modeling will assess associations between treatment and objective response.
Duration of response | From the time a response is experienced to progression or death, assessed up to 3 years
Incidence of, causality, and outcome of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will described using National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. Will be summarized with descriptive statistics: mean, median, standard deviation, minimum, and maximum for continuous variables, and frequencies and percentages for categorical variables.
Incidence of, causality, and outcome of serious AEs | Up to 30 days after last dose of study treatment
  AEs will be assessed as defined by NCI-CTCAE v 5.0. Will be summarized with descriptive statistics: mean, median, standard deviation, minimum, and maximum for continuous variables, and frequencies and percentages for categorical variables.
Changes in vital signs and laboratory values | Up to 30 days after last dose of study treatment
  Will be summarized with descriptive statistics: mean, median, standard deviation, minimum, and maximum for continuous variables, and frequencies and percentages for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, Principal Investigator — City of Hope Medical Center
Locations (13):
- United States (13):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope at Newport Beach Fashion Island, Newport Beach, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - City of Hope at Chicago, Zion, Illinois